CLINICAL TRIAL: NCT01777776
Title: A Phase Ib/II, Multicenter, Study of LEE011 in Combination With LGX818 in Adult Patients With BRAF Mutant Melanoma.
Brief Title: Safety and Efficacy of LEE011 and LGX818 in Patients With BRAF Mutant Melanoma.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to scientific and business considerations.
Sponsor: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X2105
Record Dates: First submitted 2013-01-22; First posted 2013-01-29 (Estimated); Results first posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-07

CONDITIONS: Locally Advanced Metastatic BRAF Mutant Melanoma
Keywords: Open-label dose escalation; BRAF inhibitor; LEE011; CDK4/6; LGX818; RAF kinase inhibitor; Metastatic melanoma; BRAF; V600
MeSH Terms: conditions — Melanoma | interventions — ribociclib; encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase Ib (Experimental): Phase Ib will randomize 18 patients with BRAF mutant melanoma, who are naïve or who have progressed on prior therapy to evaluate the safety and tolerability of the combination of LEE011 and LGX818.
  Interventions: Drug: LEE011; Drug: LGX818
- Phase II arm 1a (Experimental): Phase II arm 1a will randomize 60 patients that are naïve to prior BRAF inhibitor therapy to LGX818+LEE011 to evaluate the effect of adding LEE011 to a BRAFi in this population.
  Interventions: Drug: LEE011; Drug: LGX818
- Phase II arm 1b (Experimental): Phase II arm 1b will randomize 30 patients to LGX818. Single agent anti-tumor activity of LGX818 is comparable to other BRAFi that are either approved or in clinical trials. This single agent anti-tumor activity will be compared to that of the combination (LEE011 + LGX818) in the BRAFi naïve patient population.
  Interventions: Drug: LGX818
- Phase II arm 2 (Experimental): Phase II arm 2 will evaluate a single arm LEE011+LGX818 in 40 patients resistant to prior BRAF inhibitor therapy. Single agent LGX818 has shown limited activity in patients with melanoma who have failed prior BRAF inhibitor treatment; the contribution of LEE011 in this combination will be evaluated.
  Interventions: Drug: LEE011; Drug: LGX818

INTERVENTIONS:
Drug: LEE011 — LEE011 will be administered orally, once daily for 21 consecutive days followed by a 7-day planned break (28-day cycle).
  Other Names: Ribociclib
  Arms: Phase II arm 1a; Phase II arm 2; Phase Ib
Drug: LGX818 — LGX818 will be administered orally, once daily on a continuous dosing schedule (28-day cycle).
  Other Names: Encorafenib

SUMMARY:
To evaluate the safety, tolerability and efficacy of LEE011 and LGX818 when administered orally to patients with BRAF mutant melanoma.

DETAILED DESCRIPTION:
In response to developments in the treatment of melanoma, the sponsor reviewed the data from the ongoing study and decided to halt further enrollment of patients in the Phase Ib part of the study. Consequently, the Phase II part of the study was not performed. Early termination of the study was not due to any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of locally advanced or metastatic melanoma along with written documentation of BRAF V600 mutation.
* ECOG performance status of 0 - 2.
* Patients enrolled into Phase Ib must have evidence of evaluable and/or measurable disease as determined by RECIST v1.1.
* Patients enrolled into Phase II (BRAFi naïve and resistant) must have evidence of measurable disease as determined by RECIST v1.1.
* Archival tumor tissue must be obtained for patients enrolled in Phase Ib and Phase II arm 1a/b- BRAFi naïve patients. If an archival tumor tissue is not available, a fresh tumor sample is acceptable.
* For patients enrolled in the phase II arm 2, patients must agree to undergo a fresh tumor biopsy unless one was collected prior to study entry but at the time of disease relapse from the most recent BRAFi treatment.

Exclusion Criteria:

* Symptomatic brain metastases.
* Symptomatic or untreated leptomeningeal disease.
* Patients with inadequate laboratory values during screening.
* In the phase II BRAFi naïve arms (1a/b), prior exposure to CDK4/6 inhibitor (e.g., PD 0332991)
* Impaired cardiac function or clinically significant cardiac diseases.
* Impairment of gastro-intestinal (GI) function or GI disease that may significantly alter the absorption of LEE011 or LGX818.
* Patients with concurrent severe and/or uncontrolled concurrent medical conditions.
* Previous or concurrent malignancy.
* Major surgery < 2 weeks before starting study treatment
* Known diagnosis of human immunodeficiency virus (HIV) or hepatitis C.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Array BioPharma, Study Director — 303-381-6604
Locations (9):
- United States (5):
  - University of Colorado Dept of Oncology, Aurora, Colorado
  - Karmanos Cancer Institute Dept of Oncology, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center Dept Oncology, New York, New York
  - Oregon Health & Science University Dept. of OHSU (3), Portland, Oregon
  - Vanderbilt University Medical Center SC - Dept of Oncology ., Nashville, Tennessee
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Woodville, South Australia
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Utrecht, Netherlands, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment to CLEE011X2105 began on 10-July-2013. The study concluded on 13-April-2015. Participant Flow data is comprised of the Full Analysis Set (FAS), which is all patients who received at least one dose of LGX818 or LEE011.
  Not completed subjects represents subjects that stopped treatment early, due to the corresponding reason.
Pre-assignment Details: In response to developments in the treatment of melanoma, the sponsor reviewed the data from the ongoing study and decided to halt further enrollment of patients in the Phase Ib part of the study. Consequently, the Phase II part of the study was not performed. Early termination of the study was not due to any safety concerns.
Groups:
- Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort); Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort); Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort); Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort): Ribociclib (LEE011) was provided in capsule form for oral use and was to be taken orally, once a day for 21 consecutive days followed by a 7-day planned break as part of each 28-day cycle of treatment.
  Encorafenib (LGX818) was to be provided in capsule form for oral use and taken orally, once a day for 28 consecutive days as part of each 28-day cycle of treatment.
Period: Overall Study
Arm/Group | Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort) | Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort)
Started | 6 | 12 | 6 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 12 | 6 | 4
Not completed — Adverse Event | 2 | 4 | 0 | 0
Not completed — Disease Progression | 4 | 8 | 6 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data is comprised of the Full Analysis Set (FAS), which is all patients who received at least one dose of LGX818 or LEE011.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort) | Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort) | Total
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 10 | 4 | 2 | 18
  >=65 years | 4 | 2 | 2 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (10.71) | 49.8 (13.66) | 58.0 (10.55) | 62.0 (17.63) | 56.6 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 1 | 0 | 11
  Male | 3 | 5 | 5 | 4 | 17
Weight [Mean (Standard Deviation); unit: kilograms] | 84.60 (12.793) | 78.08 (17.069) | 80.17 (10.308) | 74.70 (16.415) | 79.44 (14.450)
WHO/ECOG performance status [Number; unit: participants] — Categories:
  * 0 - Fully active, able to carry on all pre-disease performance without restriction
  * 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * 2 - Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  * 3 - Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  * 4 - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  participants
    0 | 2 | 4 | 1 | 1 | 8
    1 | 4 | 7 | 5 | 3 | 19
    2 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib - Incidence of Dose Limiting Toxicities (DLTs) in Cycle 1
Description: Dose Limiting Toxicities (DLTs) during the first 28 days of the combination treatment of LEE011 and LGX818.
  Due to the halt of enrollment, no Maximum Tolerated Dose (MTD) was formally declared during the study.
Time Frame: Cycle 1 (approximately 28 days)
Population: Analysis group is comprised of the Safety Set (SS), which includes all patients who received at least one dose of LEE011 or LGX818, and have at least one valid post-baseline safety assessment.
Measure: Number; unit: participants with DLTs
Arm/Group | Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort) | Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort)
Number analyzed (Participants) | 6 | 12 | 6 | 4
participants with DLTs
  Myalagia | 1 | 0 | 0 | 0
  Elevated Bilirubin | 1 | 0 | 0 | 0
  Neuralgia | 0 | 0 | 1 | 0
  Maculopapular Rash | 0 | 0 | 0 | 1

2. Primary Outcome: Phase II - Progression Free Survival (PFS)
Description: As per RECIST v1.1, PFS is the time from date of randomization/ start of treatment to the date of event defined as the first documented progression or death due to any cause.
  Due to the halt of enrollment during the Phase Ib part of the study, all analyses related to efficacy were not performed.
Time Frame: Approximately 23 months after enrollment
Population: This analysis set would have been the Full Analysis (FAS), which included all patients who received at least one dose of encorafenib or ribociclib.
Groups:
- Phase II - Arm 1a (LGX818+LEE011): Patients naïve to prior BRAF inhibitor therapy were administered LGX818+LEE011 to evaluate the effect of adding LEE011 to a BRAFi in this population.
  LEE011: Administered orally, once daily for 21 consecutive days followed by a 7-day planned break (28-day cycle).
  LGX818: Administered orally, once daily on a continuous dosing schedule (28-day cycle).
- Phase II - Arm 1b (LGX818): Patients administered LGX818. Single agent anti-tumor activity of LGX818 is comparable to other BRAFi that are either approved or in clinical trials. This single agent anti-tumor activity will be compared to that of the combination (LEE011 + LGX818) in the BRAFi naïve patient population.
  LGX818: Administered orally, once daily on a continuous dosing schedule (28-day cycle).
Arm/Group | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Phase II - Objective Response Rate (ORR)
Description: As per RECIST v1.1, ORR is defined as the proportion of patients with a best overall response of complete response or partial response.
  Due to the halt of enrollment during the Phase Ib part of the study, all analyses related to efficacy were not performed.
Time Frame: Approximately 23 months after enrollment
Population: as for outcome 2
Groups:
- Phase II - Arm 2 (BRAFi Resistant): Patients with BRAF V600 mutant melanoma who are resistant to selective BRAFi treatment will be enrolled into LEE011+ LGX818.
Arm/Group | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase I - Number of Subjects Experiencing at Least One Adverse Event (AE).
Time Frame: Approximately 23 months after enrollment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort) | Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort)
Number analyzed (Participants) | 6 | 12 | 6 | 4
participants | 6 | 12 | 6 | 4

5. Secondary Outcome: Phase I - Number of Subjects Experiencing at Least One Serious Adverse Event (SAE).
Time Frame: Approximately 23 months after enrollment
Population: Analysis group is comprised of the Safety Set (SS), which is all patients who received at least one dose of LEE011 or LGX818, and have at least one valid post-baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort) | Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort)
Number analyzed (Participants) | 6 | 12 | 6 | 4
participants | 3 | 5 | 3 | 1

6. Secondary Outcome: Phase Ib/II - Plasma Concentration-time Profiles
Description: Due to the halt of enrollment during the Phase Ib part of the study, all analyses related to plasma concentration time profiles were not performed.
Time Frame: 28-day cycles
Population: This analysis group would have been the PK analysis set (PAS), which would have consisted of all patients who had at least one blood sample providing evaluable drug concentration data.
Groups:
- Phase I (Dose Escalation): Adult patients with locally advanced or metastatic BRAF V600 mutant melanoma who are resistant to selective BRAFi treatment or patients who are naïve to selective BRAFi treatment.
  LEE011: Administered orally, once daily for 21 consecutive days followed by a 7-day planned break (28-day cycle).
  LGX818: Administered orally, once daily on a continuous dosing schedule (28-day cycle).
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Phase Ib/II - Overall Response Rate (ORR)
Description: ORR is defined as the proportion of patients with a best overall response of complete response or partial response.
  Due to the halt of enrollment during the Phase Ib part of the study, this analysis was not performed.
Time Frame: Approximately 23 months after enrollment
Population: as for outcome 2
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Phase Ib/II - Progression Free Survival (PFS)
Description: PFS is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause.
  Due to the halt of enrollment during the Phase Ib part of the study, this analysis was not performed.
Time Frame: Approximately 23 months after enrollment
Population: as for outcome 2
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase Ib/II - Duration Of Response (DOR)
Description: DOR is calculated as the time from the date of first documented response (complete response (CR) or partial response (PR)) to the first documented date of progression or death due to underlying cancer.
  Due to the halt of enrollment during the Phase Ib part of the study, this analysis was not performed.
Time Frame: Approximately 23 months after enrollment
Population: as for outcome 2
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Phase II - Overall Survival (OS)
Description: OS is defined as the time from date of randomization/start of treatment to date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last known date patient alive.
  Due to the halt of enrollment during the Phase Ib part of the study, this analysis was not performed.
Time Frame: Approximately 23 months after enrollment
Population: as for outcome 2
Arm/Group | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Phase Ib/II - Pharmacokinetic Parameters: AUCtau
Description: Due to the halt of enrollment during the Phase Ib part of the study, all analyses related to pharmacokinetic parameters were not performed.
Time Frame: 28-day cycles
Population: as for outcome 6
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Phase Ib/II - Pharmacokinetic Parameters: Cmin
Description: as for outcome 11
Time Frame: 28-day cycles
Population: as for outcome 6
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Phase Ib/II - Pharmacokinetic Parameters: Cmax
Description: as for outcome 11
Time Frame: 28-day cycles
Population: as for outcome 6
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Phase Ib/II - Pharmacokinetic Parameters: Tmax
Description: as for outcome 11
Time Frame: 28-day cycles
Population: as for outcome 6
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Phase Ib/II - Pharmacokinetic Parameters: Racc
Description: as for outcome 11
Time Frame: 28-day cycles
Population: as for outcome 6
Arm/Group | Phase I (Dose Escalation) | Phase II - Arm 1a (LGX818+LEE011) | Phase II - Arm 1b (LGX818) | Phase II - Arm 2 (BRAFi Resistant)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: This study began recruitment on 10-July-2013 and concluded on 13-April-2015. Adverse Events (AEs) were collected throughout the study, approximately 2 years.
Description: An AE is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after patient's signed informed consent has been obtained.
Arm/Group | Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort) | Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort) | Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort)
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/12 | 3/6 | 1/4
Other Adverse Events (participants affected / at risk) | 6/6 | 12/12 | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort) (N=6) | Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort) (N=12) | Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort) (N=6) | Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort) (N=4)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall abscess (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Simple partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: LEE011 200 mg + LGX818 300 mg (Cohort) (N=6) | Phase Ib: LEE011 300 mg + LGX818 200 mg (Cohort) (N=12) | Phase Ib: LEE011 400 mg + LGX818 100 mg (Cohort) (N=6) | Phase Ib: LEE011 400 mg + LGX818 200 mg (Cohort) (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 6 (6) | 4 (4) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xerosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin sensitisation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ephelides (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study recruitment was halted on 07-Aug-2014 during the Phase Ib part of the study. The Phase II part of the study was not performed. Early termination of the study was not due to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of the sponsor's agreements with its investigators may vary. However, the sponsor does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in the clinical trial.